CLINICAL TRIAL: NCT02261129
Title: Bioequivalence of the 80 mg Telmisartan Film-coated Tablet Compared With Two Tablets of the Conventional 40 mg Telmisartan Tablet Following Oral Administration in Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Two-sequence, Four-period Replicated Crossover Study)
Brief Title: Bioequivalence of Telmisartan Film-coated Tablet Compared With Two Tablets of the Conventional Telmisartan Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.557
Record Dates: First submitted 2014-10-09; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- Telmisartan, film-coated tablet (Experimental): one tablet of telmisartan
  Interventions: Drug: Telmisartan film-coated tablet
- Telmisartan, conventional tablet (Active Comparator): Two tablets of telmisartan
  Interventions: Drug: Telmisartan uncoated tablet

INTERVENTIONS:
Drug: Telmisartan film-coated tablet
  Arms: Telmisartan, film-coated tablet
Drug: Telmisartan uncoated tablet
  Arms: Telmisartan, conventional tablet

SUMMARY:
Study to demonstrate the bioequivalence of the telmisartan 80 mg film-coated tablet vs. two tablets of the telmisartan 40 mg conventional tablet

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (Blood pressure, pulse rate, body temperature), 12-lead ECG, clinical laboratory tests
   * 1.1 No findings deviating from normal and of clinical relevance
   * 1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥20 and ≤35 years
3. Body weight≥50kg
4. Body Mass Index ≥18.0 and ≤25.0 kg/m2
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate, body temperature, and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. Chronic or relevant acute infections
6. History of relevant allergy/hypersensitivity (including allergy to a drug or its excipients)
7. Any clinical relevant findings of the laboratory test deviating from normal
8. Positive result for either hepatitis B antigen, anti hepatitis C virus antibodies, syphilitic test or human immunodeficiency virus (HIV) test
9. History of surgery of gastrointestinal tract (except appendectomy)
10. History of relevant orthostatic hypotension (mean standing systolic blood pressure (SBP) varies by ≥20 mmHg from mean supine SBP or mean standing diastolic blood pressure (DBP) varies by ≥10 mmHg from mean supine DBP), fainting spells or blackouts
11. History of hepatic dysfunction (e.g. biliary cirrhosis, cholestasis)
12. History of serious renal dysfunction
13. History of bilateral renal artery stenosis or renal artery stenosis in a solitary kidney
14. History of cerebrovascular disorder
15. History of hyperkalemia
16. Known hypersensitivity to any component of the telmisartan formulation, or to any other angiotensin II receptor blockers
17. Intake of drugs with a long half-life (≥24 hours) within at least one month or less than 10 half-lives of the respective drug before administration of the investigational product
18. Use of any drugs within 10 days before administration of the investigational product or during the trial
19. Participation in another trial with an investigational drug within four months before administration of the investigational product or during the trial
20. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
21. Alcohol abuse
22. Drug abuse
23. Blood donation (100 mL or more) within four weeks before administration of the investigational product
24. Excessive physical activities within one week before administration of the investigational product or during the trial
25. Intake of alcohol within 2 days prior to administration
26. Inability to comply with dietary regimen of study centre
27. Inability to refrain from smoking on trial days
28. Any other clinical conditions that investigator or sub-investigator judges that the subject is ineligible for study participation

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to last quantifiable data point (AUC0-tz) | up to 72 hours after drug administration
Maximum measured concentration of the analyte in plasma (Cmax) | up to 72 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 72 hours after drug administration
Time from dosing to the maximum measured concentration of the analyte in plasma (tmax) | up to 72 hours after drug administration
Terminal rate constant of the analyte in plasma (λz) | up to 72 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 72 hours after drug administration
mean residence time of the analyte in the body after po administration (MRTpo) | up to 72 hours after drug administration
Number of subjects with adverse events | up to 72 hours after last drug administration